CLINICAL TRIAL: NCT04956952
Title: Enhanced External Counterpulsation in Patients With Fontan Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Fred Wu, MD, Principal Investigator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P00037795
Record Dates: First submitted 2021-06-01; First posted 2021-07-09 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Single-ventricle; Congenital Heart Disease
Keywords: Fontan
MeSH Terms: conditions — Univentricular Heart; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Enhanced External Counterpulsation (EECP) (Other): 1 hour of treatment with EECP
  Interventions: Device: EECP

INTERVENTIONS:
Device: EECP — 1 hour of treatment with EECP

SUMMARY:
The purpose of the proposed study is to determine the safety of enhanced external counterpulsation (EECP), a system for compressing the blood vessels in the legs in synchrony with an individual's cardiac rhythm, in clinically well, adult Fontan patients, to document the acute hemodynamic and myocardial effects of EECP on the Fontan circulation, and to demonstrate acute changes in endothelial function after one hour of the procedure.

DETAILED DESCRIPTION:
The investigators plan to study the effects of enhanced external counterpulsation (EECP), on patients who have had Fontan surgery for treatment of complex congenital heart disease. Eligible patient volunteers will undergo a series of biophysical measurements at rest including echocardiographic assessment of ventricular function, pulmonary blood flow/cardiac output measurement using an inert gas rebreathing method (Innocor), and measurements of biomarkers of endothelial function (ET-1, NOx). Patients will then undergo 1 hour of treatment with EECP, during which additional echocardiographic assessment of ventricular function and pulmonary blood flow/cardiac output measurements will be performed at multiple levels of leg compression. Subjects will be assessed periodically for adverse effects and discomfort during the EECP treatment. At the completion of treatment, patients will be allowed 30 minutes to rest before undergoing one more echocardiographic assessment of ventricular function, pulmonary blood flow/cardiac output measurement, and measurements of biomarkers of endothelial function (ET-1, NOx). Measurements made during and after treatment will be compared to baseline measurements.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Fontan physiology being seen in the Boston Children's Hospital cardiology clinic for outpatient care.

Exclusion Criteria:

* Current pregnancy
* Decompensated heart failure/pulmonary edema
* Severe aortic insufficiency
* Active tachyarrhythmias
* Frequent atrial or ventricular ectopy
* Symptomatic peripheral vascular disease
* Thrombophlebitis or history of deep vein thrombosis or stasis ulcer
* Aortic aneurysm
* Uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure>110 mmHg)
* Systolic blood pressure <90 mmHg
* Active femoral site bleeding or hematoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Change in cardiac output | Immediately prior to starting EECP treatment, during each 20-minute phase of EECP treatment, and 30 minutes after EECP treatment
  Measurement of cardiac output (pulmonary blood flow) in L/min using inert gas rebreathing method (Innocor CO device)
Total number and type of adverse events during EECP treatment | During EECP treatment (duration 60 minutes)
  Adverse events will be collected by an investigator and documented using CTCAE criteria
Total number and type of adverse events immediately following EECP treatment | From completion of EECP treatment until patient discharge (30 to 60 minutes)
  Adverse events will be collected by an investigator and documented using CTCAE criteria

SECONDARY OUTCOMES:
Change in ventricular strain analysis | Immediately prior to starting EECP treatment, during each 20-minute phase of EECP treatment, and 30 minutes after EECP treatment
  Global mid-ventricle circumferential strain (%) and global longitudinal strain (%) calculated from speckle-tracking echocardiography
Change in qualitative ventricular systolic function | Immediately prior to starting EECP treatment, during each 20-minute phase of EECP treatment, and 30 minutes after EECP treatment
  Qualitative assessment of systolic function of dominant ventricle on 2-dimensional echocardiography, categorized as normal, low normal to mildly depressed, mildly depressed, mildly to moderately depressed, moderately depressed, moderately to severely depressed, severely depressed, or unable to determine.
plasma endothelin (ET-1) | pre and 30 minutes post EECP treatment
  This will measure endothelial function
Total nitrate/nitrite (NOx) levels | pre and 30 minutes post EECP treatment
  This will measure endothelial function

CONTACTS AND LOCATIONS:
Overall Officials: Fred Wu, MD, Principal Investigator — Attending Cardiologist
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No